CLINICAL TRIAL: NCT01703884
Title: Improved Quality of ANC and Diagnostic Services for Malaria in Pregnancy
Brief Title: ANC & Malaria Diagnostic in Pregnancy
Acronym: AQUAMOD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Muraz (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Tinto Halidou, PharmD, Msc, PhD, Centre Muraz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B00531
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Malaria
Keywords: Malria diagnosis; Malaria prevention in pregnancy; ANC services improvement
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASAQ (Experimental): In the intervention area, obstetric, medical, drug-exposure histories will be collected at ANC visits. In addition, in the last trimester of the pregnancy women will be systematically evaluated with RDT for whether they have malaria parasites and treated effectively.
  Interventions: Drug: ASAQ
- SP (No Intervention): At ANC and labor wards for women in the control area, there will be no change from routine approaches.

INTERVENTIONS:
Drug: ASAQ — In the intervention area, obstetric, medical, drug-exposure histories will be collected at ANC visits. In addition, in the last trimester of the pregnancy (> 28 weeks of pregnancy), women will be systematically evaluated with malaria RDT for whether they have malaria parasites and treated effectively with ASAQ.
  Other Names: Coarsucam, ASAQ Winthrop
  Arms: ASAQ

SUMMARY:
The program's overall objective is to assess the impact of a package of interventions aimed at reducing malaria-related mortality and morbidity in pregnant women and newborns by ensuring access to a package of interventions designed to optimise the detection and treatment of malaria during pregnancy as well as improving the early detection and treatment of malaria during the third trimester.

DETAILED DESCRIPTION:
This is a cluster-randomised study in which the health facility is the unit of randomisation. 16 health facilities will be randomised to intervention and control. At the community level women will be encouraged to access ANC early in the pregnancy, attend follow-up antenatal visits throughout the pregnancy and deliver at the facility. The current recommended standard of care will be provided to all women attending antenatal and obstetric care. In the intervention area, obstetric, medical, drug-exposure histories will be collected at ANC visits. In addition, in the last trimester of the pregnancy (> 28 weeks of pregnancy), women will be systematically evaluated with selected diagnostic test for whether they have malaria parasites and treated effectively. Skilled birth attendants at the facility will be trained in emergency obstetric and neonatal care and the assessment of neonates for danger signs, low birth weight and external/observable birth defects. In the control area, women will be provided with standard practice of care. In both areas, women will be diagnosed and treated at delivery if they are positive.

ELIGIBILITY:
Inclusion Criteria:

* Located in the geographical location of Dafra & Do district
* Have a minimum attendance of 200 pregnant women per year

Exclusion Criteria:

* other public health facilities, private clinics and Dafra District Hospital will be excluded from the study.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5254 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Placental malaria at delivery | 9 months
  The main outcome variable of interest will be the proportion of women in each group with placental malaria at delivery (defined as placental biopsies positive for P. falciparum )

SECONDARY OUTCOMES:
The proportion of women with peripheral positive malaria infection at delivery | 9 months
  The proportion of women with peripheral positive malaria infection at delivery (defined via detection of asexual stages of P. f alciparum by microscopy)

OTHER OUTCOMES:
The proportion of women with severe anaemia in women at delivery | 9 months
  The proportion of women with severe anaemia in women at delivery (severe anaemia defined as Hg <8 g/dL),
Low Birth Weight | 9 months
  Low Birth Weight (defined as <2500g)
Stillbirth | 28 weeks of gestation
  Stillbirth (defined as dead birth after 28 weeks of gestation)
Perinatal and early neonatal deaths | 7 days post delivery
  Perinatal and early neonatal deaths (i.e. death within 7 days of birth)
External/observable birth defects | 9 months
  Presence of external/observable birth defects in neonates identified at birth or as soon as possible thereafter.
Maternal death | 42 days post delivery
  Maternal death (death within 42 days of delivery, regardless of cause)

CONTACTS AND LOCATIONS:
Overall Officials: Halidou Tinto, PharmD, PhD, Principal Investigator — centre muraz - irss
Locations (1):
- Dafra & Do districts, Bobo-Dioulasso, Hauts Bassins-houet, Burkina Faso